CLINICAL TRIAL: NCT01412242
Title: Identification of the Optimal Approach to the Ultrasound Diagnosis of Deep Vein Thrombosis of the Lower Extremities in Symptomatic Patients
Brief Title: Simplification of the Diagnosis of Deep Vein Thrombosis
Acronym: PALLADIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Paolo Prandoni, Professor of Internal Medicine, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2188P
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep vein thrombosis; Ultrasonography; Pulmonary embolism; D-dimer; Pre-test probability
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extensive search for isolated calf DVT (Experimental): As this is a prospective cohort study, for definition there is only 1 arm
  Interventions: Other: Extensive search for isolated calf DVT

INTERVENTIONS:
Other: Extensive search for isolated calf DVT — Extensive search for isolated calf DVT in patients with negative CUS of the proximal veins who have a high PTP and a positive D-dimer

SUMMARY:
Prospective cohort study aimed at simplifying the diagnostic approach to symptomatic patients with the clinical suspicion of deep vein thrombosis (DVT) of the lower extremities. All patients will receive a pre-test clinical probability (PTP) and the determination of D-dimer. Patients with low PTP and negative D-dimer will have the diagnosis ruled out. All other patients will undergo compression ultrasonography (CUS) of the proximal vein system. Patients with negative CUS and either low PTP or negative D-dimer will have the diagnosis ruled out, while those with high PTP and positive D-dimer will undergo extensive ultrasound investigation of the calf vein system. All patients in whom the diagnosis of DVT is ruled out will be followed-up prospectively up to three months for documenting the development of symptomatic thromboembolic events.

DETAILED DESCRIPTION:
All eligible patients will undergo D-dimer measurement and a formal assessment of pre-test clinical probability (PTP) by means of the Wells score. Patients with unlikely PTP and negative D-dimer will have DVT ruled out and will undergo a 3-month clinical follow-up. If at least one of the two tests is positive, patients will undergo CUS of the proximal vein system by investigating at least the common femoral vein at the groin, the superficial femoral vein at the mid thigh and the popliteal vein(s) in the popliteal fossa. A positive CUS will adjudicate proximal DVT. In the case of negative CUS of the proximal vein system, patients with either negative D-dimer or unlikely PTP will have DVT ruled out, and will undergo a 3-month follow up. Only patients with concomitant likely PTP and positive D-dimer will undergo whole-leg ultrasonography with interrogation of the calf veins. A positive test will adjudicate distal DVT. Patients with negative test will undergo a 3-month clinical follow up.

Follow-up. All patients in whom DVT is ruled out will be monitored for 3 months (either by clinical visit or by telephone contact) after the enrolment in the study. Patients with clinical symptoms of DVT or PE during follow-up will undergo objective diagnostic testing (venous ultrasound for suspected DVT and spiral CT-scan or VQ scan for suspected PE). All source documents will be sent out for an independent adjudication. In case of death, PE diagnosis will be adjudicated by means of autopsy, if available. If autopsy is not available, the adjudication of PE-related death will be done based on clinical documentation.

D-dimer. All quantitative D-dimer tests available at each center will be acceptable for the purpose of this study. D-dimer will be considered negative according to the cut-offs provided by manufacturers.

Sample size. The investigators expect that in every 100 symptomatic outpatients DVT will be excluded without the need for objective testing in approximately 30%, while approximately 20% will have a CUS-detected proximal DVT, approximately 15% will have negative CUS and unlikely PTP in spite of positive D-Dimer (no need for further investigation), approximately 15% will have negative CUS and negative D-Dimer in spite of likely PTP (no need for further investigation, and approximately 20% will have negative CUS and both likely PTP and positive D-Dimer (thus requiring interrogation of the calf vein system).

The investigators hypothesize that the incidence of venous thromboembolic events during follow up in patients labeled as not having DVT will not exceed 1% with the application of the proposed algorithm, and that the upper limit of the 95% confidence intervals around this proportion will not exceed 2%. Accordingly, ap proximately 1100 patients should be enroled.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with clinically suspected DVT
* signed informed consent

Exclusion Criteria:

* concomitant signs or symptoms of pulmonary embolism
* previous DVT of the affected leg
* referral for superficial vein thrombosis or bilateral DVT
* ongoing or planned anticoagulant therapy
* need for pharmacological thromboprophylaxis (e.g. recent surgery or medical disease)
* inpatient status
* unavailability to follow up
* pregnancy
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Safety of withdrawing anticoagulation from patients labeled as not having DVT on the basis of a one-day examination | Up to 3 months
  To assess the rate of symptomatic thromboembolic events occurring up to 3 months after DVT exclusion

SECONDARY OUTCOMES:
The rate of isolated calf vein thrombi | Up to 1 day
  Patients with high PTP and positive D-dimer in spite of negative CUS of the proximal vein system will undergo extensive search for isolated calf vein DVT.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Prandoni, MD, PhD, Study Chair — University of Padua, Italy
Locations (1):
- Paolo Prandoni, Padua, Italy

REFERENCES:
- [Derived] Ageno W, Camporese G, Riva N, Iotti M, Bucherini E, Righini M, Kamphuisen PW, Verhamme P, Douketis JD, Tonello C, Prandoni P; PALLADIO Study Investigators. Analysis of an algorithm incorporating limited and whole-leg assessment of the deep venous system in symptomatic outpatients with suspected deep-vein thrombosis (PALLADIO): a prospective, multicentre, cohort study. Lancet Haematol. 2015 Nov;2(11):e474-80. doi: 10.1016/S2352-3026(15)00190-8. Epub 2015 Oct 18. PMID 26686257